CLINICAL TRIAL: NCT04121611
Title: Optical Coherence Tomography Guided Antithrombotic Treatment After Endovascular Thrombectomy of the Posterior Circulation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Dr. Victor Yang, Neurosurgeon, Sunnybrook Health Sciences Centre
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1192019
Record Dates: First submitted 2019-10-08; First posted 2019-10-10 (Actual); Last update posted 2019-10-17 (Actual); Status verified 2019-10

CONDITIONS: Stroke of Basilar Artery; Optical Coherence Tomography; Antithrombotics; Endovascular Thrombectomy
Keywords: Basilar; Stroke; Thrombus; Optical Coherence Tomography
MeSH Terms: conditions — Stroke; Thrombosis | interventions — Heparin; Aspirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Optical coherence tomography confirmed residual thrombus (Experimental): Early antithrombotics
  Interventions: Drug: Unfractionated heparin; Drug: Acetylsalicylic Acid (ASA)
- Optical coherence tomography confirmed no residual thrombus (No Intervention): Best medical management

INTERVENTIONS:
Drug: Unfractionated heparin — 1. Intravenous unfractionated heparin (UFH) infusion within 6 hours of EVT with target activated partial thromboplastin time (aPTT) 64-86
  2. Anticoagulation to continue for minimum of 48 hours (can be maintained on UFH aPTT 64-86 or transitioned to low-molecular weight heparin (LMWH) Enoxaparin 1mg/kg)
  Arms: Optical coherence tomography confirmed residual thrombus
Drug: Acetylsalicylic Acid (ASA) — 1. Acetylsalicylic Acid (ASA) 325mg PO/PR/NG loading dose < 2 hours of EVT completion
  2. ASA 81mg PO OD maintenance dose
  Arms: Optical coherence tomography confirmed residual thrombus

SUMMARY:
Evidence regarding the role of early (<24 hours) antithrombotics post-revascularization with either intravenous thrombolysis (IVT), endovascular thrombectomy (EVT), or a combination of both remains scarce. In 2018 the American Heart Association/American Stroke Association changed their recommendation, stating that the risk of antithrombotic therapy within the first 24 hours after treatment with IVT (with or without EVT) is uncertain. This was changed after data emerged that early antithrombotics may be safe and may improve outcomes in select patients undergoing EVT.

Recently the investigators showed for the first time that significant residual basilar thrombus can exist after EVT despite complete angiographic revascularization using endovascular optical coherence tomography imaging. This residual thrombus could cause ongoing function-limiting strokes with occlusion of vital basilar perforators after EVT. Therefore, the investigators propose a prospective,non-randomized safety study to evaluate optical coherence tomography guided antithrombotic management for patients with confirmed residual thrombus after EVT for basilar occlusion.

ELIGIBILITY:
Inclusion Criteria:

- All patients deemed candidates for endovascular thrombectomy(EVT) for basilar artery occlusion. As no robust guidelines exist for the role of EVT in patients with acute basilar artery occlusion, the decision for EVT is made by a team of stroke neurologist and neuro-interventionalist at our regional stroke center.

Exclusion Criteria:

* High-density lesion consistent with hemorrhage of any degree.
* Significant established infarct size.
* Contraindication to receiving post-revascularization antithrombotics for any reason (history of major hemorrhage in the past six months, hereditary or acquired bleeding diathesis, major surgery within last three months, platelets <100 X 109 /L, coagulation factor deficiency, already on anticoagulant that would not allow administration of UFH)
* Informed consent is not or cannot be obtained.
* Females of childbearing potential who are known to be pregnant and/or lactating or who have positive pregnancy tests on admission.
* Other serious, advanced, or terminal illness.
* Patients who require hemodialysis or peritoneal dialysis.
* Uncontrolled hypertension defined as systolic blood pressure>185 mm Hg or diastolic blood pressure>110mm Hg that cannot be controlled except with continuous parenteral antihypertensive medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2019-10-14 (Actual); Primary Completion 2021-10-14 (Estimated); Study Completion 2021-12-14 (Estimated)

PRIMARY OUTCOMES:
Favorable outcome | 90 days
  Favorable outcome at day 90 defined as a modified Rankin Score (mRS - functional scale) of 0-3.

SECONDARY OUTCOMES:
Symptomatic Intracranial Hemorrhage | 24 hours CT imaging ± 8 hours.
Incidence of residual thrombus | Immediately after endovascular thrombectomy
  Fraction of patients with residual thrombus after endovascular thrombectomy as observed with optical coherence tomography
Excellent Outcome | 90 days
  Excellent outcome at day 90 defined as a modified Rankin Score (mRS - functional scale) of 0-2.

CONTACTS AND LOCATIONS:
Locations (1):
- Sunnybrook Heath Sciences Center, Toronto, Ontario, Canada

REFERENCES:
- [Background] Pasarikovski CR, Ramjist J, da Costa L, Black SE, Yang V. Optical coherence tomography imaging after endovascular thrombectomy for basilar artery occlusion: report of 3 cases. J Neurosurg. 2019 Aug 23;133(4):1141-1146. doi: 10.3171/2019.5.JNS191252. Print 2020 Oct 1. PMID 31443067
- [Background] Powers WJ, Rabinstein AA, Ackerson T, Adeoye OM, Bambakidis NC, Becker K, Biller J, Brown M, Demaerschalk BM, Hoh B, Jauch EC, Kidwell CS, Leslie-Mazwi TM, Ovbiagele B, Scott PA, Sheth KN, Southerland AM, Summers DV, Tirschwell DL; American Heart Association Stroke Council. 2018 Guidelines for the Early Management of Patients With Acute Ischemic Stroke: A Guideline for Healthcare Professionals From the American Heart Association/American Stroke Association. Stroke. 2018 Mar;49(3):e46-e110. doi: 10.1161/STR.0000000000000158. Epub 2018 Jan 24. PMID 29367334
- [Background] Schonewille WJ, Wijman CA, Michel P, Rueckert CM, Weimar C, Mattle HP, Engelter ST, Tanne D, Muir KW, Molina CA, Thijs V, Audebert H, Pfefferkorn T, Szabo K, Lindsberg PJ, de Freitas G, Kappelle LJ, Algra A; BASICS study group. Treatment and outcomes of acute basilar artery occlusion in the Basilar Artery International Cooperation Study (BASICS): a prospective registry study. Lancet Neurol. 2009 Aug;8(8):724-30. doi: 10.1016/S1474-4422(09)70173-5. Epub 2009 Jul 3. PMID 19577962
- [Background] Jeong HG, Kim BJ, Yang MH, Han MK, Bae HJ, Lee SH. Stroke outcomes with use of antithrombotics within 24 hours after recanalization treatment. Neurology. 2016 Sep 6;87(10):996-1002. doi: 10.1212/WNL.0000000000003083. Epub 2016 Aug 12. PMID 27521435